CLINICAL TRIAL: NCT07296965
Title: The Role of the Oral Microbiome in Carotid Atherosclerosis: Investigating in a Cross-sectional Study the Microbial Influence on Plaque Development and Vulnerability Based on Biobank Data
Brief Title: Oral Microbiome in Carotid Atherosclerosis
Acronym: OMICA
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: National Research, Development and Innovation Office, Hungary (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sótonyi Péter, MD, DSc, Head of Department of Vascular and Endovascular Surgery, Semmelweis University Heart and Vascular Center
Other Study IDs: NKFI-Advanced 149634; NKFI-Advanced 149634 (Other Grant/Funding Number: National Research, Development, and Innovation Office); BM/33955-1/2023 (Other: Semmelweis University Carotid Plaque Biobank)
Record Dates: First submitted 2025-11-24; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerosis Cardiovascular Disease; Atherosclerosis of Artery; Carotid Artery Plaque; Periodontitis; Carotid Artery Diseases
Keywords: Oral Microbiome; Carotid Plaque; Plaque vulnerability; Atherosclerosis; Periodontal disease; Biobank study; Microbial colonization
MeSH Terms: conditions — Carotid Stenosis; Periodontitis; Carotid Artery Diseases; Atherosclerosis; Periodontal Diseases; Communicable Diseases | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Oral swabs, anal swabs, urine samples, blood samples, and carotid plaque tissue obtained during carotid endarterectomy will be retained. Samples will be stored in the Semmelweis University Carotid Plaque Biobank (BM/33955-1/2023). DNA will be extracted for microbiome analysis using next-generation sequencing and may also be used for confirmatory molecular assays. All biospecimens will be de-identified and stored under controlled conditions for future research on vascular and microbial interactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vulnerable Plaque Group: Participants with vulnerable carotid plaques, identified based on ultrasound gray-scale median (GSM) score, photon-counting CT angiography, and MR plaque characterization.
  Interventions: Other: Sample Collection
- Stable Plaque Group: Participants with stable carotid plaques, classified by imaging criteria indicating low vulnerability.
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — Participants undergo preoperative oral health evaluation and the collection of oral, anal, urine, blood, and carotid plaque samples during carotid endarterectomy for microbiome analysis. All samples are fully anonymized and processed within the Semmelweis University Carotid Plaque Biobank (BM/33955-1/2023). No experimental treatments are administered; all activities occur within the framework of biobank-approved surgical and diagnostic procedures.
  Other Names: Oral-Systemic Microbiome Analysis; Carotid Plaque Microbiome Sampling

SUMMARY:
The goal of this observational study, called OMICA (Oral Microbiome in Carotid Atherosclerosis), is to learn how bacteria living in the mouth may influence the development and stability of plaques in the carotid arteries, which supply blood to the brain. Plaque buildup in these arteries can lead to stroke.

Researchers want to understand whether certain oral bacteria are linked to plaque vulnerability, meaning a higher chance that the plaque will rupture and cause a stroke.

The study will include a cohort of adults scheduled for carotid endarterectomy at Semmelweis University. Participants will be enrolled in the Semmelweis University Carotid Biobank project.

The main questions the study aims to answer are:

Do people with more severe gum disease or tooth infection have a higher number of bacteria in their carotid plaques, and are those plaques more likely to rupture?

Are the bacteria found in vulnerable plaques different from those in stable plaques?

Are similar bacteria found in the mouth, gut, and plaques, suggesting that bacteria may travel through the body?

What participants will do:

Have their oral health checked before surgery, including an exam of gum disease and tooth infections.

Provide microbiome samples from the mouth, anus, urine, and carotid plaque (taken during surgery).

Have preoperative photon-counting computed tomography (CT) performed to assess plaque stability and study eligibility.

All samples and imaging data will be analyzed to identify bacterial species and their relationship to plaque type.

The study does not involve any experimental treatment or medication. Participation adds no significant medical risk beyond standard care.

Researchers will compare bacterial patterns between people with vulnerable plaques and those with stable plaques to identify microbial signatures linked to carotid plaque instability.

The results may help create future microbiome-based risk models for detecting people at higher risk of stroke or severe atherosclerosis.

DETAILED DESCRIPTION:
Background and Rationale: Cardiovascular diseases are currently the leading cause of death globally, according to the World Health Organization. Recent studies report a 4.2% prevalence of moderate to severe carotid artery stenosis. A growing body of evidence highlights the association between poor oral health and vascular disease. Periodontitis is a highly prevalent condition, affecting approximately 10% of the global population with its severe form (1). Several studies have revealed correlations between the severity of periodontal disease and the presence of pathogenic bacteria in carotid (2) and atherosclerotic plaques (3).

Methods:

Population: The cross-sectional study includes a cohort of patients undergoing carotid endarterectomy: roughly half with vulnerable and half with stable carotid plaques. Photon-counting computed tomography (CTA) is part of the preoperative eligibility assessment confirming internal carotid artery stenosis and determining inclusion in the study. Only non-invasive magnetic resonance (MR) and ultrasound imaging will be requested from participants as part of the study protocol for classification of plaque vulnerability. All imaging data will be anonymized in accordance with Semmelweis University data protection protocols.

Intervention (Sample Collection): This study involves preoperative oral health evaluation and the collection of oral, anal, urine, blood, and carotid plaque samples during carotid endarterectomy for microbiome analysis. All samples and corresponding data will be fully anonymized and processed within the Semmelweis University Carotid Plaque Biobank (BM/33955-1/2023).

Comparator: Patients with vulnerable vs. stable carotid plaques, as classified by carotid duplex ultrasound (GSM score) and photon-counting CTA and MR plaque characterization.

Outcome:

1. Identification of periodontal and endodontic pathogens in the oral microbiome that positively correlate with plaque severity and vulnerability.
2. Distinct microbiome compositions in carotid plaques of patients with stable versus vulnerable lesions, supporting the role of bacterial colonization in plaque instability.
3. Detection of microbiome similarities across oral, anal, and vascular samples, suggesting systemic bacterial dissemination that may contribute to carotid stenosis progression.

Expected Value of Results: This project integrates microbiome and imaging data to explore links between oral bacteria and carotid plaque vulnerability. By investigating the interplay between oral microbiota and vascular disease, the study aims to deepen our understanding of plaque pathogenesis and progression. The findings may contribute to developing microbiome-based risk prediction models for plaque vulnerability, supported by advanced imaging data.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed internal carotid artery (ICA) stenosis on preoperative photon-counting computed tomography (CTA)
* Adults (≥18 years) undergoing carotid endarterectomy at Semmelweis University.
* Eligible for surgery based on standard anesthesiologic evaluation.
* Willing and able to provide written informed consent for participation and sample collection.

Exclusion Criteria:

* Active systemic infection or current antibiotic therapy within 30 days before surgery.
* Immunosuppressive therapy or immunodeficiency disorders.
* Inability to undergo MRI (e.g., pacemaker, metallic implants, severe claustrophobia).
* Pregnancy or lactation.
* Malignancy under active treatment.
* Prior carotid surgery or stenting on the same side.
* Refusal or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients undergoing carotid endarterectomy at Semmelweis University, Budapest, Hungary, within the framework of the Semmelweis Carotid Plaque Biobank. Eligible individuals are adults with confirmed internal carotid artery stenosis identified by photon-counting CT angiography. Enrollment is consecutive among surgical candidates who provide informed consent. The study population reflects a tertiary vascular surgery center cohort representing both stable and vulnerable plaque phenotypes, as classified by ultrasound, MR, and CTA imaging.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Identification of Oral and Carotid Plaque Microbiome Associations | At time of carotid endarterectomy
  Microbiome composition of oral and carotid plaque samples will be analyzed using next-generation sequencing to identify bacterial taxa correlated with plaque vulnerability. Relative abundance and diversity indices will be compared between participants with vulnerable and stable carotid plaques to determine microbial associations linked to plaque instability.

SECONDARY OUTCOMES:
Differences in Microbiome Composition Between Vulnerable and Stable Carotid Plaques | At time of carotid endarterectomy
  Microbial diversity, relative abundance, and taxonomic composition of carotid plaque samples will be compared between vulnerable and stable plaques using 16S rRNA gene sequencing and bioinformatic analysis. Results will help identify microbial signatures associated with plaque stability or vulnerability.
Identification of Shared Microbial Taxa Across Oral, Anal, Urine, and Carotid Plaque Samples | At time of carotid endarterectomy
  Microbiome overlap among oral, anal, urine, and carotid plaque samples will be analyzed to detect bacterial species present across multiple body sites, indicating possible systemic dissemination pathways linked to atherosclerotic plaque progression.

OTHER OUTCOMES:
Correlation Between Oral Health Status and Carotid Plaque Vulnerability | Within 2 weeks prior to carotid endarterectomy
  Clinical periodontal indices (probing depth, attachment loss, and periapical lesion presence) will be correlated with imaging-defined plaque vulnerability scores to evaluate whether oral disease severity predicts plaque instability.

CONTACTS AND LOCATIONS:
Locations (1):
- Városmajor Heart and Vascular Center, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be de-identified and may be shared with qualified researchers upon reasonable request following completion of the study and publication of primary results, pending ethical and institutional approval.

REFERENCES:
- [Background] Isoshima D, Yamashiro K, Matsunaga K, Taniguchi M, Matsubara T, Tomida S, Ota S, Sato M, Shimoe Y, Kohriyama T, Arias Z, Omori K, Yamamoto T, Takashiba S. Microbiome composition comparison in oral and atherosclerotic plaque from patients with and without periodontitis. Odontology. 2021 Jan;109(1):239-249. doi: 10.1007/s10266-020-00524-w. Epub 2020 May 19. PMID 32430725
- [Background] Brun A, Nuzzo A, Prouvost B, Diallo D, Hamdan S, Meseguer E, Guidoux C, Lavallee P, Amarenco P, Leseche G, Bouchard P, Michel JB, Range H. Oral microbiota and atherothrombotic carotid plaque vulnerability in periodontitis patients. A cross-sectional study. J Periodontal Res. 2021 Apr;56(2):339-350. doi: 10.1111/jre.12826. Epub 2020 Dec 25. PMID 33368263
- [Background] Frencken JE, Sharma P, Stenhouse L, Green D, Laverty D, Dietrich T. Global epidemiology of dental caries and severe periodontitis - a comprehensive review. J Clin Periodontol. 2017 Mar;44 Suppl 18:S94-S105. doi: 10.1111/jcpe.12677. PMID 28266116
- See also: Biobank — https://semmelweis.hu/research/services/biobank/
- See also: Városmajor Biobank - Transplant Biobank — https://semmelweis.hu/biobank/biobankok/varosmajori-biobank-transzplantacios-biobank/

DOCUMENTS (2):
  • Informed Consent Form: Consent Form (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT07296965/ICF_000.pdf
  • Informed Consent Form: Information Form (2025-05-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT07296965/ICF_001.pdf